CLINICAL TRIAL: NCT03680820
Title: Pediatric Gastroparesis Registry: Pediatric Registry of Patients With Suspected Gastroparesis
Brief Title: Pediatric Gastroparesis Registry
Acronym: PGpR
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Baylor College of Medicine (Other); Nationwide Children's Hospital (Other); Boston Children's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Other Study IDs: 8 DK PGpR; U01DK112194 (NIH); U24DK074008 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-09-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis; Gastroparesis-like Syndrome
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, peripheral blood mononuclear cells (PBMC), GI mucosal biopsies (in those undergoing upper GI endoscopy), urine, and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ages 5-9, gastroparesis: Participants 5-9 years of age at screening with documented gastroparesis (delayed gastric emptying)
- Ages 5-9, gastroparesis-like syndrome: Participants 5-9 years of age at screening with cardinal symptoms of gastroparesis, but who have normal gastric emptying
- Ages 10-17, gastroparesis: Participants 10-17 years of age at screening with documented gastroparesis (delayed gastric emptying)
- Ages 10-17, gastroparesis-like syndrome: Participants 10-17 years of age at screening with cardinal symptoms of gastroparesis, but who have normal gastric emptying

SUMMARY:
The objective of the Pediatric Gastroparesis Registry is to create a national prospective registry of children and adolescents with gastroparesis and gastroparesis-like syndrome (symptoms of gastroparesis but normal gastric emptying).

DETAILED DESCRIPTION:
In the Pediatric Gastroparesis Registry (PGpR), we will collect detailed epidemiological, clinical, psychological, and patient outcome data with the goal of classifying patients with gastroparesis and gastroparesis-like syndromes into pathophysiologically defined phenotypes.

The Primary Objective is to create a national prospective registry of children and adolescents with gastroparesis and gastroparesis-like syndrome (symptoms of gastroparesis but normal gastric emptying) to include:

1. Demographic, clinical, psychological, nutritional characteristics, physiological measures, and serial assessments of symptoms over 3 years while receiving clinical care;
2. Establish a Biorepository of plasma, serum, peripheral blood mononuclear cells (PBMC), GI mucosal biopsies (in those undergoing upper GI endoscopy), urine and stool collected from the children and adolescents in this registry which will allow for future analyses such as cytokines, bacterial DNA and microbiome to investigate the etiology and pathogenesis of gastroparesis in children.

Secondary Objectives:

1. To determine what factors, if any, play a role in the outcomes of children who do not improve within two years of diagnosis
2. To assess the spectrum of symptom severity of the cardinal gastroparesis symptoms: nausea, vomiting, early satiety, postprandial fullness (and upper abdominal pain, if present) in children with gastroparesis
3. To assess several areas of gastric motility in pediatric patients with symptoms of gastroparesis (e.g., intragastric meal distribution, global gastric emptying)
4. To capture the clinical symptomatic course (outcome) of pediatric patients followed in the registry
5. To determine whether gastroparesis symptoms are correlated with gastric emptying in a pediatric population
6. To characterize abdominal pain in patients with gastroparesis and gastroparesis-like syndrome by using questionnaires, water load satiety testing and quantitative sensory testing (QST)
7. Determine the prevalence of hypermobility spectrum disorders in pediatric patients with gastroparesis
8. To determine if the volume of water consumed during the water load satiety test is an indirect measure of gastric accommodation
9. To determine if the water load satiety test is associated with an increased severity of gastroparesis symptoms (fullness, bloating, abdominal pain, etc).
10. To compare the intragastric meal distribution during scintigraphy to symptoms of early satiety, postprandial fullness in patients with symptoms of gastroparesis
11. Define immune cell profiles, cytokine induction and epigenetic changes in diabetic and idiopathic gastroparesis

ELIGIBILITY:
Inclusion Criteria:

* Cardinal symptoms of gastroparesis of at least 12 weeks duration. Cardinal symptoms of gastroparesis are the constellation of some combination of: nausea, vomiting, early satiety, postprandial fullness; symptoms sometimes may be accompanied by upper abdominal pain
* An etiology of either diabetic, idiopathic, or post-fundoplication gastroparesis or gastroparesis-like disorder (symptoms of gastroparesis but normal gastric emptying; see below)
* Gastric emptying scintigraphy (GES) of solids using the 4-hour Egg Beaters® protocol (or equivalent generic liquid egg white meal) within the last 12 months with either:

  1. Abnormal gastric emptying rate defined as an abnormal 2-hour (>60% retention) and/or 4-hour (>10% retention) result based on a 4-hour scintigraphic gastric emptying study. (This group will comprise ~75% of patients in the registry)
  2. Patients with a normal gastric emptying rate, but who have symptoms of gastroparesis. (This group will comprise ~25% of patients in the registry)
* Age at least 5 years, and under 18 years at initial screening visit

Exclusion Criteria:

* Inability to comply with or complete the scintigraphic gastric emptying test (including allergy to eggs)
* Pregnancy
* Autism spectrum disorder, significant developmental delay, psychosis, or a history of bipolar disorder (because of inability to complete the gastroparesis symptom questionnaires: 24-hour recall and gastroparesis cardinal symptom questionnaire (the latter to be completed during the scintigraphy if possible)
* Use of narcotic analgesics greater than three days per week
* Presence of conditions associated with GI mucosal disease (e.g., inflammatory bowel disease, known eosinophilic gastroenteritis or eosinophilic esophagitis)
* Presence of any other condition that could cause delayed gastric emptying including:

  1. Gastrointestinal obstruction confirmed by EGD, UGI, or abdominal CT
  2. Primary neurological conditions that can cause nausea and vomiting such as increased intracranial pressure, space occupying or inflammatory/infectious lesions
  3. Acute or chronic renal failure (abnormal creatinine for age) and/or on hemodialysis or peritoneal dialysis
  4. Acute liver failure
  5. Advanced liver disease (features of portal hypertension)
* Clinically significant congenital heart disease (i.e., vagal injury during cardiac repair)
* History of esophageal, gastric or bowel surgery excepting prior fundoplication
* Metabolic disease including mitochondrial disease and inborn errors of metabolism
* Chronic lung disease (including cystic fibrosis)
* A serious chronic medical condition (e.g., cystic fibrosis)
* Use of medications that can affect motility during the gastric emptying study
* Any other condition, which in the opinion of the investigator, could explain the symptoms or interfere with study requirements
* Inability to obtain informed consent/assent

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 5-9 yrs. of age [n=210] and 10-17 yrs. of age [n=210] suspected of having gastroparesis at the time they are undergoing gastric scintigraphy or who have undergone scintigraphy in the past 12 months with documented gastroparesis or gastroparesis-like syndrome (symptoms of gastroparesis but normal gastric emptying; 25% of the proposed study number 105 out of 420).
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in water load satiety volume consumed | 24 weeks
  The Water Load Satiety Test involves the participant drinking refrigerated spring water (4 degrees C) from a 1-liter container over a period of 5 minutes until feeling completely full. The total volume of water consumed (mL) over 5 minutes is the unit of measure, and the outcome is assessed by calculating the change in volume consumed (24 weeks - baseline).

SECONDARY OUTCOMES:
Change in Pediatric Quality of Life (PedQL) Generic Core Scale | 48 weeks
  Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale is completed by the child, and is composed of 23 items comprising 4 dimensions: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Each item is answered using a 3-point scale: 0 (Not at all), 2 (Sometimes), 4 (A lot). Items are reversed scored and linearly transformed to a scale from 0 to 100, with higher scores indicating lower problems. The Total Score is calculated as the sum of all the items over the number of items answered on all the scales. The outcome is assessed by calculating the change in Total Score (48 weeks - baseline).
Change in Pediatric Quality of Life (PedQL) Gastrointestinal Symptom Scale | 48 weeks
  Pediatric Quality of Life (PedQL) Gastrointestinal Symptoms Scale is completed by the child, and is composed of 58 items comprising 10 dimensions: Stomach Pain and Hurt, Stomach Discomfort When Eating, Food and Drink Limits, Trouble Swallowing, Heart Burn and Reflux, Nausea and Vomiting, Gas and Bloating, Constipation, Blood in Poop, and Diarrhea. Each item is answered using a 3-point scale: 0 (Not at all), 2 (Sometimes), 4 (A lot). Items are reversed scored and linearly transformed to a scale from 0 to 100, with higher scores indicating lower problems. The Symptom Total Scales Score is calculated as the sum of the items answered in the 10 dimensions. The outcome is assessed by calculating the change in Total Score (48 weeks - baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Shulman, MD, Study Chair — Baylor College of Medicine
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Public use complete database will be submitted to the NIDDK Data Repository
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: By the end of the funding period.
Access Criteria: Application through NIDDK Data Repository; IRB approval
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: Study website — https://jhuccs1.us/gpcrc/